CLINICAL TRIAL: NCT06906224
Title: Effects of Different Doses of Buspirone Combined With Clozapine on Psychiatric Symptoms and Cognitive Function in Patients With Schizophrenia: A Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Buspirone Combined With Clozapine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chuanfu Song (Other)
Collaborators: Wuhu Fourth People's Hospital affiliated with Bengbu Medical University (Other)
Responsible Party: Sponsor-Investigator, Chuanfu Song, Director, Wuhu Fourth People's Hospital affiliated with Bengbu Medical University
Organization: Wuhu Fourth People's Hospital affiliated with Bengbu Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wuhu4thPeopleH001
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: Buspirone; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Control Groups; Clozapine; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): Patients received oral clozapine (Jiangsu Pharmaceutical Co., Ltd., Approval No. H32022963) in combination with a placebo. Each dose of the placebo was 1 mg, taken three times a day. Use of placebo: This study employed a double-blind design. Patients in the control group received clozapine monotherapy and took a placebo concurrently. The placebo was identical to buspirone tablets in terms of appearance, shape, colour and packaging to guarantee the double-blind nature of the study. The placebo was custom-made by a third-party pharmaceutical company. Its label only stated 'placebo' and was exactly the same as that of buspirone tablets. This design was intended to eliminate the potential impact of the placebo effect on the study results.
  Interventions: Drug: Control group (clozapine, placebo)
- Low-dose group (Active Comparator): Patients received oral buspirone tablets (Jiangsu Enhua Pharmaceutical Co., Ltd., Approval No. H19991024) in combination with clozapine. The total daily dose of buspirone was 15 mg, divided into three administrations. The dose remained unchanged throughout the entire study period.
  Interventions: Drug: Low-dose group (buspirone tablets, clozapine)
- High-dose group (Experimental): Patients received oral buspirone tablets in combination with clozapine. The initial total daily dose of buspirone was 15 mg, divided into three administrations. One week later, the dose was increased to a total daily dose of 30 mg, also divided into three administrations.
  Interventions: Drug: High-dose group (buspirone tablets, clozapine)

INTERVENTIONS:
Drug: Control group (clozapine, placebo) — Patients received oral clozapine (Jiangsu Pharmaceutical Co., Ltd., Approval No. H32022963) in combination with a placebo. Each dose of the placebo was 1 mg, taken three times a day.
  Arms: Control group
Drug: Low-dose group (buspirone tablets, clozapine) — Patients received oral buspirone tablets (Jiangsu Enhua Pharmaceutical Co., Ltd., Approval No. H19991024) in combination with clozapine. The total daily dose of buspirone was 15 mg, divided into three administrations. The dose remained unchanged throughout the entire study period.
  Arms: Low-dose group
Drug: High-dose group (buspirone tablets, clozapine) — Patients received oral buspirone tablets in combination with clozapine. The initial total daily dose of buspirone was 15 mg, divided into three administrations. One week later, the dose was increased to a total daily dose of 30 mg, also divided into three administrations.
  Arms: High-dose group

SUMMARY:
This study aimed to evaluate the enhancing effects of different doses of buspirone on psychiatric symptoms and cognitive function in patients with schizophrenia. The investigators adopted a prospective, randomised, double-blind, placebo-controlled study design and included 46 patients with schizophrenia being treated at the Fourth People's Hospital of Wuhu. The patients were randomly divided into three groups: the control group, the low-dose group and the high-dose group. The control group received clozapine monotherapy, while the experimental groups received additional buspirone at different doses in addition to clozapine. The Positive and Negative Syndrome Scale (PANSS) and the Chinese version of the Repeatable Battery for the Assessment of Neuropsychological Status were used to evaluate psychiatric symptoms and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years;
* Meeting the diagnostic criteria for chronic schizophrenia in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Current remission of psychotic symptoms. The patients had a relatively stable mental state in the past 4 weeks, with a total score of ≤60 points and a score of ≤4 points on the Positive and Negative Syndrome Scale (PANSS)[15], and there were no signs of acute psychotic symptoms. To ensure that patients were included in the chronic phase, only patients who had been diagnosed with schizophrenia for ≥1 year were recruited, thus avoiding confusion with acute phase cases;
* Receiving monotherapy with antipsychotic drugs, such as clozapine.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients allergic to buspirone;
* Patients previously diagnosed with cognitive impairment, such as dementia or intellectual disability;
* Patients with a history of other brain injuries or diseases, such as stroke, traumatic brain injury, epilepsy or intracranial infection;
* Patients with severe liver or kidney insufficiency;
* Patients with severe physical diseases or other mental illnesses, such as bipolar disorder, major depressive disorder, alcohol or substance dependence;
* Patients with a history of using drugs that affect cognitive function during the study period or those who need to adjust the existing treatment regimen;
* Patients who are unable to cooperate with cognitive function tests or have poor treatment compliance.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of psychiatric symptoms | 4 weeks, 8 weeks and 12 weeks
  The PANSS was used to evaluate the severity of psychiatric symptoms in schizophrenia. The PANSS is composed of three subscales: Positive Scale, Negative Scale and General Psychopathology Scale. Each item is rated on a scale from 1 to 7, with a total score ranging from 0 to 125; lower scores indicate milder symptoms.
Assessment of cognitive function | 4 weeks, 8 weeks and 12 weeks
  Cognitive function was assessed using the Chinese version of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)[17]. The RBANS assesses five cognitive domains: immediate memory, visuospatial/constructional abilities, language, attention and delayed memory. Each domain contains specific tasks and scoring criteria.
Adverse event records | 4 weeks, 8 weeks and 12 weeks
  Throughout the entire study period, detailed records were made of all adverse events reported by patients, including the type of the event, the occurrence time, the duration and the severity level. Particular attention was paid to the potential adverse reactions associated with the combined use of medications, such as drowsiness and dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhu Fourth People's Hospital affiliated with Bengbu Medical University, Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No